CLINICAL TRIAL: NCT00570167
Title: Comparison of Hip Resurfacing and Cementless Metal-on-metal Total Hip Arthroplasty - Prospective Randomized Clinival Trial
Brief Title: Comparison of Hip Resurfacing and Cementless Metal-on-metal Total Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Kuopio University Hospital (Other); University of Turku (Other)
Responsible Party: Ville Remes, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TYH7306; ISRCTN60907614
Record Dates: First submitted 2007-12-05; First posted 2007-12-10 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Hip Osteoarthritis
Keywords: Osteoarthritis; Hip; Artroplasty; Resurfacing
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Active Comparator): Total cementless hip arthroplasty with metal-on-metal bearings
  Interventions: Procedure: Cementless total hip arthroplasty with m-o-m bearings
- 1 (Active Comparator): Hip resurfacing
  Interventions: Procedure: Hip resurfacacing

INTERVENTIONS:
Procedure: Hip resurfacacing — Hip resurfacing with cementless acetabular cup and cemented femoral head
  Other Names: BHR (Smith & Nephew, Memphis, TN, USA)
  Arms: 1
Procedure: Cementless total hip arthroplasty with m-o-m bearings — Cementless monoblock acetabular cup and cementless femoral stem with modular large head and metal-on-metal bearings..
  Other Names: BHR-cup and Synergy stem (Smith & Nephew. Memphis, TN, USA)
  Arms: 2

SUMMARY:
To compare clinical, functional and radiological outcome after hip resurfacing and cementless metal-on-metal total hip arthroplasty.

DETAILED DESCRIPTION:
While many problems associated with endoprosthetic surgery have been solved, there are still some open questions: In hip replacement one of the most controversial issues is the role and the indications for "resurfacing" (Schmalzried 2005, Hungerford 2005).

Resurfacing In traditional hip replacement, the head of the femur is replaced with a metal head secured to a stem in the femoral canal. In hip resurfacing, the neck of the femur is not cut, and instead the head of the femur is capped with a hemispherical metal ball articulated with an acetabular cup. The concept of resurfacing was developed as early as the 1970s, but it was abandoned due to unsatisfactory results. The procedure started to spark new interest in the 1990s as the results improved due to improvements in the articulation surfaces and fixation techniques (Amstutz 1998), and it has become considerably more common in the 2000s. In Australia, for example, resurfacing procedures accounted for 9% of all hip replacement operations carried out as a consequence of primary osteoarthritis, and their use has increased 17-fold in the 2000s (Australian Orthopedic Association National Joint Replacement Registry).

The partly assumed benefits of hip resurfacing include less bone resection in connection with the procedure, easiness of reoperation (a "conventional" replacement is carried out if reoperation is necessary), smaller risk of dislocation due to the larger head, and more physiological flexibility of the femur as the neck of the femur is not replaced with an inflexible metal stem. The short-term and mid-term results of modern resurfacing procedures presented in the reports of the developer clinics have been encouraging (Daniel 2004, Beaule 2004), but long-term results are lacking. Resurfacing procedures are technically more challenging and have given rise to complications that are not associated with conventional hip replacement, such as fractures of the femoral neck (Shimmin 2005). On the other hand, the socket and the diameter of the ball used in resurfacing procedures and conventional hip replacements are similar, and excellent results have been reached with modern conventional cementless stems (Eskelinen 2005). There are no published studies comparing modern resurfacing prostheses to solutions involving cementless stems with a large head and metal-on-metal articulation surfaces.

ELIGIBILITY:
Inclusion Criteria:

1. Primary osteoarthritis of the hip, planned to be treated by hip replacement surgery
2. Normal acetabulum, or no more than mild dysplasia of the acetabulum
3. Aged 18 to 60 years
4. The patient's mother tongue is Finnish

Exclusion Criteria:

1. Patient has a secondary osteoarthritis of hip
2. The patient has undergone endoprosthetic surgery of the other hip in the preceding six months, or such a procedure is planned for the patient in the next six months
3. The patient has undergone or is planned to undergo endoprosthetic surgery of the knee or ankle in the next year
4. The patient has undergone surgery of the other hip, knee or ankle with an unsatisfactory outcome
5. The patient has been diagnosed with or is suspected to have an untreated or recurring malignancy or systemic infection
6. A disease treated with cortisone or immunosuppressive medication
7. The patient's cooperation is impaired for any reason
8. Any systemic disease that impairs the patient's mobility
9. Female patients in fertile age who are planning to have children during the study
10. The patient has previously undergone an operation of the hip region that extended below the subcutaneous tissue
11. The patient has experienced a femoral neck fracture
12. The patient has been diagnosed with or is strongly suspected to have osteoporosis (T-score less than or equal to -2.5 SD)
13. The patient has a systemic or metabolic disease that has impaired or is going to impair bone quality
14. A significant cyst (diameter greater than 1 cm) or cysts in the area of the femoral neck
15. Bilateral simultaneous hip arthroplasty
16. Neck-shaft angle 120 degrees or less
17. Deformed femoral head making hip resurfacing impossible
18. Head-neck ratio less than 1.2
19. Avascular necrosis of the femoral head

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Estimated)
Dates: Start 2006-11

PRIMARY OUTCOMES:
Pain and discomfort on Visual Analogue Score (VAS) scale and in 7-point Likert-scale. | At 2, 5 and 10 years

SECONDARY OUTCOMES:
A difference of 15 points in WOMAC questionnaire | At 2, 5 and 10 years
Difference in 20-metre walking test and 3-metre "up and go" test | At 2, 5 and 10 years
Difference in the observed change in the quality of life | At 2, 5 and 10 years
Difference in the observed cost-effectiveness | At 2, 5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ville M Remes, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (3):
- Finland (3):
  - Kuopio University Hospital, Kuopio, Itä-Suomi
  - Turku University Hospital, Turku, Lounais-Suomi
  - Helsinki University Hospital, Helsinki, Uusimaa